CLINICAL TRIAL: NCT04411576
Title: Studies on Current and Past SARS-CoV-2 Infection (and COVID-19) in Healthcare in Stockholm, Sweden
Brief Title: Current and Past SARS-CoV-2 Infection and COVID-19 in Healthcare
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Dillner, Professor of Infectious Disease Epidemiology; Director of R&D, Karolinska University Hospital
Other Study IDs: COVID-19 Studien
Record Dates: First submitted 2020-05-26; First posted 2020-06-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV 2
Keywords: Healthcare; Personnel; Screening; Virus; Antibodies; Sick leave; COVID-19
MeSH Terms: conditions — Virus Diseases; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The throat samples and serum samples collected in this study will be biobanked. Information on biobanking is included in the informed consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Throat swab sample for measuring current infection with SARS-CoV-2 — Throat sample taken by the study participant to be analyzed with RT PCR for the presence of SARS-CoV-2 viral nucleic acids.
Diagnostic Test: Blood sample for serology to measure past infection with SARS-CoV-2 — Blood samples for serology to be analyzed for the presence of SARS-CoV-2 antibodies.

SUMMARY:
The SARS-CoV-2 pandemic and resulting COVID-19 disease causes a substantial burden on healthcare systems. Little is known about how the infection spreads within healthcare. In order to design control strategies, knowledge of the presence of viral nucleic acid and whether an immune response to the virus has been mounted is needed. The purpose of this study is to determine whether personnel and patients/clients in healthcare in Region Stockholm have a currrent SARS-CoV-2 infection or have had an infection. This information will be used to understand how the infection spreads in healthcare, to explore the association with sick-leave among personnel, and to plan high-quality and safe care.

Healthcare providers and organizations participating in the study from the greater Stockholm region include the following: Karolinska University Laboratory, Karolinska University Hospital; Intensive Care Unit, Karolinska University Hospital; SciLifeLab; KTH Royal Institute of Technology; Roo Home Healthcare Services (Roo Hemtjänst och Vård); Health Care Services Stockholm County (SLSO); Region Stockholm; Southern Hospital (Södersjukhuset); Danderyd Hospital; Capio St Göran Hospital; Södertälje Hospital; Tiohundra AB; Ersta Hospital, Sweden; and St Eriks Eye Hospital (St Eriks Ögonsjukhus).

ELIGIBILITY:
Inclusion Criteria (all three criteria must be fulfilled):

* Healthcare personnel or patient/client of healthcare in Stockholm County
* Age 18-99
* Provided consent to participate in the study

Exclusion Criteria:

* No informed consent to participate provided
* Already confirmed with SARS-CoV-2 infection
* Already sampled for SARS-CoV-2 infection based on clinical presention but where the result has not been reported yet

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthcare personnel, patients, and clients of healthcare in Stockholm County who do not have a confirmed or suspected SARS-CoV-2 infection form the study population and are eligible for inclusion if they fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 26326 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | Throat and blood samples are taken one time at enrollment. Other background characteristics are determined using linkages to healthcare employment databases up to two months after enrollment.
  Ongoing and past SARS-CoV-2 infection, measured in throat samples (current infection) and serum (past infection, antibodies to SARS-CoV-2) evaluated in relation to age, gender, sickleave, address, workplace, sampling date, work tasks (for healthcare personnel) and evaluated in relation to date of hospitalization, diagnoses, and interventions for patients and healthcare clients.

OTHER OUTCOMES:
SARS-CoV-2 sequencing | Sequencing will be completed in a later phase of the study, after enrollment is complete and within 1 year.
  Sequencing will be completed on the positive samples to determine is the virus isolate is the same. This can provide information on the spread of the infection in population.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
We have yet to determine whether the IPD will be available for other researchers.

REFERENCES:
- [Derived] Dillner J, Elfstrom KM, Blomqvist J, Eklund C, Lagheden C, Nordqvist-Kleppe S, Hellstrom C, Olofsson J, Andersson E, Jernbom Falk A, Bergstrom S, Hultin E, Pin E, Manberg A, Nilsson P, Hedhammar M, Hober S, Mattsson J, Muhr LSA, Conneryd Lundgren K. Antibodies to SARS-CoV-2 and risk of past or future sick leave. Sci Rep. 2021 Mar 4;11(1):5160. doi: 10.1038/s41598-021-84356-w. PMID 33664279
- [Derived] Dillner J, Elfstrom KM, Blomqvist J, Engstrand L, Uhlen M, Eklund C, Boulund F, Lagheden C, Hamsten M, Nordqvist-Kleppe S, Seifert M, Hellstrom C, Olofsson J, Andersson E, Falk AJ, Bergstrom S, Hultin E, Pin E, Pimenoff VN, Hassan S, Manberg A, Nilsson P, Hedhammar M, Hober S, Mattsson J, Arroyo Muhr LS, Lundgren KC. High Amounts of SARS-CoV-2 Precede Sickness Among Asymptomatic Health Care Workers. J Infect Dis. 2021 Jul 2;224(1):14-20. doi: 10.1093/infdis/jiab099. PMID 33580261